CLINICAL TRIAL: NCT03231111
Title: The Effectiveness of Using Preventive Multimedia Teaching Program in Lung Cancer Women Receiving Targeted Therapy on Skin-Related Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201703118RINB
Record Dates: First submitted 2017-07-13; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional group (No Intervention)
- Multimedia group (Experimental)
  Interventions: Other: Preventive Multimedia Teaching Program

INTERVENTIONS:
Other: Preventive Multimedia Teaching Program — Preventive Multimedia Teaching Program
  Arms: Multimedia group

SUMMARY:
The Effectiveness of Using Preventive Multimedia Teaching Program in Lung Cancer Women Receiving Targeted Therapy on Skin-Related Quality of Life

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 20 years of age.
2. The first time to accept the target drug treatment (Iressa, Tarceva) treatment, diagnosis of lung cancer third or fourth stage of the women.
3. There are computer equipment at home to play the disc.
4. can speak, write, read Chinese, clear consciousness, no cognitive impairment.
5. In the medical center of Taipei, a medical department, medical or surgical clinic for treatment.

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-25 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
skindex-29 | average of 1 month
  Skin-Related Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan